CLINICAL TRIAL: NCT01127490
Title: Duloxetine(Cymbalta) for Fibromyalgia: An Open-Label Pilot Study to Assess Potential Mechanisms for Fibromyalgia in Peripheral Tissue Innervation That Could Predict Therapeutic Responsiveness to Duloxetine
Brief Title: Study to Assess Mechanisms in Peripheral Tissue Innervation for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Charles Argoff, MD, Albany Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DUL2009-FFMS
Record Dates: First submitted 2010-05-18; First posted 2010-05-21 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Duloxetine — Subjects will be titrated onto Duloxetine over one week by taking 30 mg every day for seven days. Week 2 the subject will begin to take 60 mg per day until the end of the study. If the subject wishes to stop taking Duloxetine, she will be given 30 mg per day for one week for down titration.
  Other Names: Cymbalta
Procedure: Skin biopsy — 3 mm skin biopsies will be obtained from the dominant trapezius and the glabrous hypothenar area of the hand
  Other Names: Punch biopsy

SUMMARY:
The purpose of this study is to examine the characteristics of the nerves and the small veins in the skin of people with fibromyalgia. The investigators will then use this information to identify possible processes in the skin that may help explain why some people feel pain relief with the study drug (duloxetine) and others do not.

Duloxetine affects certain chemicals in the brain called neurotransmitters. An abnormality in these chemicals is thought to be related to fibromyalgia. Duloxetine is a selective serotonin and norepinephrine reuptake inhibitor (SNRI), similar to some drugs used for the treatment of depression. Duloxetine is approved for sale in the United States by the Food and Drug Administration (FDA) for the treatment of fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18-70
* Fulfill the ACR criteria for FMS (wide spread pain for at least 3 months and pain in at least 11 of 18 tender point sites.
* VAS score greater than 40mm at Screening and Randomization Visits

Exclusion Criteria:

* History of clinically significant liver disease, serious peripheral vascular disease, a blood clotting disorder, or any other medical condition felt to be exclusionary by the investigator
* Allergy to lidocaine
* Unwillingness to sign informed consent or any other reasons for which the investigator feels the subject cannot complete the study.
* Women who are pregnant, breastfeeding or trying to become pregnant
* Active cancer within the previous two years except treated basal cell carcinoma of the skin
* Presence of dermatological or neurological condition that could interfere with the interpretation of the skin biopsy or QST
* Co-existing conditions that can produce chronic widespread pain
* Presence of uncontrolled or severe depression
* Patients with pending Worker's Compensation, worker's Compensation, any ongoing litigation or disability claims due to fibromyalgia or any other source of pain, or currently receiving monetary compensation as a result of any of the above.
* Presence of uncontrolled narrow-angle glaucoma

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05-05 (Actual); Primary Completion 2015-09-09 (Actual); Study Completion 2015-09-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of duloxetine will be determined by neurological and pain assessments. | 9 weeks
  Patients will be evaluated prior to being started on duloxetine and again at eight weeks. We will use data from VAS scores, sleep diaries and quantative sensory testing.

CONTACTS AND LOCATIONS:
Overall Officials: James P. Wymer, MD, Principal Investigator — Albany Medical College
Locations (1):
- Neurosciences Institute, Albany Medical College, Albany, New York, United States